CLINICAL TRIAL: NCT00900159
Title: Effects of Daytime Eszopiclone Administration in Shift Workers on Overnight Wakefulness During a Subsequent Simulated Nightshift
Brief Title: Effects of Daytime Eszopiclone Administration in Shift Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Orfeu M. Buxton, Dr. Orfeu Buxton, Ph.D., Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ESRC-977; 2009-P-000019 (Other: Brigham and Women's Hospital)
Record Dates: First submitted 2009-04-13; First posted 2009-05-12 (Estimated); Results first posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-07

CONDITIONS: Shift-Work Sleep Disorder
Keywords: Shift-work; SWSD; eszopiclone; MWT; shiftworkers
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- eszopiclone (Experimental): Treatment with eszopiclone
  Interventions: Drug: eszopiclone
- matching placebo (Placebo Comparator): Treatment with matching placebo
  Interventions: Drug: eszopiclone; Drug: matching placebo

INTERVENTIONS:
Drug: eszopiclone — 3mg eszopiclone prior to daytime sleep for 3 days (at home) and 1 day (in lab)
  Other Names: Lunesta
Drug: matching placebo — matching placebo prior to daytime sleep for 3 days (at home) and 1 day (in lab)
  Other Names: placebo
  Arms: matching placebo

SUMMARY:
The purpose of this study is to test the effects of eszopiclone on daytime sleep and overnight wakefulness in shift workers.

DETAILED DESCRIPTION:
The current study seeks to extend the currently available treatments for SWSD by addressing the putative root cause of the problem-the inability of night-shift workers with or without SWSD- to obtain adequate daytime sleep in the face of the circadian drive for alertness that increases across the biological day. Even healthy, young subjects who are sleep-deprived overnight exhibit daytime sleep marked by frequent awakenings and low sleep efficiency, less slow-wave sleep, and altered sleep architecture, e.g. earlier predominance of REM sleep. Many night-workers routinely report 3-6 hours of habitual sleep duration for daytime sleep. Pharmacological interventions to decrease awakenings and improve total sleep time during daytime sleep could improve subsequent alertness during a night shift. Improving the wakefulness of night-shift workers over the nighttime could result in substantial benefits for the individual workers, improve workplace productivity and safety, and improve public health.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-50 (men or women)
* Current shift worker (for at least 3 months, at least 5 overnights/month and 3 consecutive)
* A willingness and ability to comply with study procedures
* If of child-bearing potential, using a medically-accepted method of birth control, including abstinence, barrier method with spermicide, steroidal contraceptive (oral, transdermal, implanted, or injected) in conjunction with a barrier method, or intrauterine device [IUD]).

Exclusion Criteria:

* Current diagnosis of DSM-IV Axis I disorder (other than insomnia)
* Regular treatment (>1time/wk) with CNS-active medication within 1 month of first inpatient visit
* Uncontrolled medical illness that would interfere with participation in the study
* BMI>32 or < 19.8 kg/m2
* Current symptoms or diagnosis of any moderate to severe sleep disorder other than SWSD
* Periodic Leg Movement of Sleep Index (PLMSi)>20/hr of sleep or Respiratory Desaturation Index (RDI)>15 on polysomnography (PSG)
* Current alcohol or drug dependence/abuse
* Menopausal or peri-menopausal symptoms that disrupt sleep
* Pregnant, lactating, or planning to become pregnant
* Current smoking of more than 10 cigarettes per day
* Current use of over the counter sleep aids such as Benadryl or melatonin

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-05; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Orfeu M Buxton, Ph.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
After publication of initial results, would require institutional data sharing agreement with Partners Inc (Brigham and Women's Hospital), and Dr. Buxton

REFERENCES:
- [Derived] Marino M, Li Y, Pencina MJ, D'Agostino RB Sr, Berkman LF, Buxton OM. Quantifying cardiometabolic risk using modifiable non-self-reported risk factors. Am J Prev Med. 2014 Aug;47(2):131-40. doi: 10.1016/j.amepre.2014.03.006. Epub 2014 Jun 17. PMID 24951039

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from April 2009 to December 2009. All recruitment happened at Brigham and Women's Hospital in Boston, MA. Recruitment included using advertisements around the Boston area.
Groups:
- Eszopiclone Then Placebo: Study participants on eszopiclone and then placebo
- Placebo Then Eszopiclone: Study participants on placebo and then eszopiclone
Period: First Intervention
Arm/Group | Eszopiclone Then Placebo | Placebo Then Eszopiclone
Started | 11 | 13
Completed | 11 | 13
Not Completed | 0 | 0
Period: Washout
Arm/Group | Eszopiclone Then Placebo | Placebo Then Eszopiclone
Started | 11 | 13
Completed | 11 | 13
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Eszopiclone Then Placebo | Placebo Then Eszopiclone
Started | 11 | 13
Completed | 10 | 13
Not Completed | 1 | 0
Not completed — disempanelled for inappropriate behavior | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eszopiclone Then Placebo | Placebo Then Eszopiclone | Total
Number analyzed (Participants) | 11 | 13 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 13 | 24
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  United States | 11 | 13 | 24

OUTCOME MEASURES:

1. Primary Outcome: Nighttime Wakefulness Assessed by Mean Sleep Latency Across 4 Maintenance of Wakefulness Tests
Description: Participants underwent four Maintenance of Wakefulness Tests (MWT) at 2-hour intervals during the simulated night shift starting 5 hours after wake time. MWT range from 0 to 40 minutes, where shorter times to fall asleep represent greater sleepiness (worse). MWT tests are averaged, for a mean in minutes.
Time Frame: On each treatment, after an 8.5 hour daytime sleep period following at least 3 consecutive night shifts
Measure: Mean (95% Confidence Interval); unit: minutes
Groups:
- Eszopiclone: Medication for insomnia symptoms
- Placebo: Non-medicated pills
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 23 | 23
minutes | 11.0 [7.5 to 22.0] | 14.75 [9.0 to 22.0]

2. Secondary Outcome: EEG-recorded Sleep Efficiency
Description: Polysomnographic recordings of daytime sleep were made at sleep screen (8.5hr) and during daytime sleep episodes of 8.5 hours of duration during treatment visits. Sleep efficiency is calculated based on the time the participant spent in bed and the actual time the participant slept.
Time Frame: On each treatment, during an 8.5-hr daytime sleep episode following at least 3 consecutive night shifts
Measure: Mean (Standard Deviation); unit: percentage of time sleeping
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 23 | 23
percentage of time sleeping | 92.3 (5.1) | 88.9 (9.6)

3. Secondary Outcome: Subjective Sleepiness and Performance
Description: The Karolinska Sleepiness Scale (KSS), a nine point Visual Analog Scale of alertness/sleepiness, was used to assess subjective sleepiness. The KSS is a scale from 1 to 9, from minimum to maximum sleepiness.
Time Frame: On each treatment, after an 8.5-hr daytime sleep episode following at least 3 consecutive night shifts
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 23 | 23
units on a scale | 5.0 (2.1) | 5.3 (2.3)

4. Secondary Outcome: Objective Vigilance Task Performance
Description: A computer-based Flanker Task elicits responses to an incongruent pairing of stimuli measured as reaction time, in milliseconds. The Flanker task tests response inhibition, or the participants suppression of an unwanted response. A target stimulus (symbol) is "flanked" by non-target stimuli (symbols) that are the same as the target stimulus, opposite of the target stimulus, or neutral with respect to the target stimulus. The task is intended to assess the ability to maintain "selective attention" in the presence of distractors.
Time Frame: On each treatment, after an 8.5 hour daytime sleep period following at least 3 consecutive night shifts
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 23 | 23
milliseconds | 631 (260.5) | 617 (294.9)

5. Secondary Outcome: Sleep-dependent Memory Consolidation
Description: A computer-based Word-pair tasks is the number of words recalled after sleep from a list of words shown prior to going to sleep.
Time Frame: On each treatment, after an 8.5 hour daytime sleep period following at least 3 consecutive night shifts
Measure: Mean (Standard Deviation); unit: words
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 23 | 23
words | 20.4 (8.1) | 21.4 (6.7)

ADVERSE EVENTS:
Description: Adverse events characterized as per clinicaltrials.gov standards. All event were "Other (Not Including Serious) Adverse Events: Adverse events that are not Serious Adverse Events. "
  Systematic methods included regular investigator assessment.
Groups:
- Placebo: eszopiclone: 3mg eszopiclone prior to daytime sleep for 3 days (at home) and 1 day (in lab)
  placebo: matching placebo prior to daytime sleep for 3 days (at home) and 1 day (in lab)
Arm/Group | Eszopiclone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 16/24 | 10/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eszopiclone (N=24) | Placebo (N=24)
Bad taste (Gastrointestinal disorders) | 10 (10) | 0 (0)
Headache (General disorders) | 6 (7) | 1 (3)
Dizziness (Cardiac disorders) | 2 (2) | 0 (0)
Nausea (General disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Somnolence (Psychiatric disorders) | 1 (2) | 2 (2)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremities (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Application site dryness (General disorders) | 0 (0) | 1 (1)
Dry eyes (Eye disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Gagging (Gastrointestinal disorders) | 0 (0) | 1 (1)
Head cold (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hunger (General disorders) | 0 (0) | 1 (1)
Leg cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Listlessness (Psychiatric disorders) | 0 (0) | 1 (1)
Short-term memory loss (Psychiatric disorders) | 0 (0) | 1 (1)
Tunnel vision (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less